CLINICAL TRIAL: NCT07007858
Title: Effects of High-Velocity Passive Stretching Protocol on Spasticity, Functional Status, and Muscle Architecture in Children With Spastic Cerebral Palsy
Brief Title: Effects of High-Velocity Passive Stretch on Spasticity, Function, and Muscle Structure in Spastic CP Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, İsa Cüce, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/197
Record Dates: First submitted 2025-05-09; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy (CP); Spastic Diplegia Cerebral Palsy; Spastic Hemiplegic Cerebral Palsy
Keywords: exercise; strecthing; muscle fascicle; ultrasound; cerebral palsy; botulinum toxin
MeSH Terms: conditions — Cerebral Palsy; Cerebral palsy, spastic, diplegic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Stretching + Standard Physical Therapy following BoNT-A Injection (Active Comparator): Participants received BoNT-A injections into the gastrocnemius muscle at clinically appropriate doses, based on individual clinical presentations and within established indications.
  In addition to standard physical therapy-including strengthening exercises, weight-bearing activities, balance training, proprioceptive exercises, and gait training-a standardized ankle joint stretching protocol was administered three sessions per week under the supervision of a physiotherapist.
  Stretching was performed for 15 minutes per leg per session, consisting of 10 repetitions of 60-second stretches with 30-second rest intervals between repetitions. The intervention period lasted four weeks. During this period, the exercises were administered by a physiotherapist. In parallel, the exercise program was taught to the families, and following the supervised phase, it was continued as a home-based exercise program for up to six months.
  Interventions: Other: Exercise
- High-Velocity Stretching + Standard Physical Therapy following BoNT-A Injection (Experimental): Participants received BoNT-A injections into the gastrocnemius muscle at clinically appropriate doses, based on their individual clinical presentation and within established indications.
  In addition to standard physical therapy-including strengthening exercises, weight-bearing activities, balance training, proprioception, and gait training-a rapid stretching protocol was administered. Rapid stretching was performed starting from the initial position, first at the slowest possible velocity (V1) for 5 minutes, as described in the Tardieu method, followed by stretching at the fastest possible velocity (V3), sufficient to elicit a catch, for 10 minutes. A 1-minute rest period was provided during each stretching session.
  This protocol was conducted three times per week for four weeks under the supervision of a physiotherapist. After the supervised phase, the stretching exercises were taught to the families and continued at home for up to six months as a home-based program, without veloci
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — In addition to standard physical therapy (including strengthening exercises, weight-bearing, balance, proprioception, and gait training), stretching will be applied to the ankle joint as described by Tardieu: first at a velocity as slow as possible (V1) for 5 minutes, followed by stretching at the fastest possible velocity (V3), sufficient to elicit a catch, for 10 minutes. A 1-minute rest period will be provided between each stretch. This protocol will be conducted three times per week for four weeks under the supervision of a physiotherapist. Afterward, the exercise will be taught to the families and continued at home as a home-based program for up to six months, without velocity measurement.
  Other Names: Standard physical therapy + High-velocity stretching
  Arms: High-Velocity Stretching + Standard Physical Therapy following BoNT-A Injection
Other: Exercise — In addition to standard physical therapy (including strengthening exercises, weight-bearing, balance, proprioception, and gait training), standard stretching will be applied to the ankle joint three sessions per week. Stretching will be performed for a total of 15 minutes per leg in each session, consisting of 10 repetitions of 60 seconds with 30-second rest intervals. During the 4-week intervention period, the exercises will be taught to the families and continued at home as a home exercise program for up to six months
  Other Names: Standard physical therapy + Standard stretching
  Arms: Standard Stretching + Standard Physical Therapy following BoNT-A Injection

SUMMARY:
One of the traditional exercises applied to cerebral palsy (CP) is passive stretching exercises. Passive stretching exercises can be applied to these patients at various speeds. A recent study has shown that high-speed passive stretching in children with CP can increase muscle bundle length in spastic muscles. Therefore, high-speed stretching exercises may potentiate the positive effects of BoNT-A treatment on spasticity and muscle fascicle in patients with CP.

This study aims to investigate whether fast stretching exercises administered to children with CP following BoNT-A injection are more effective than standard stretching in improving spasticity, functional status, and muscle architecture.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is characterized as a neurodevelopmental disorder resulting in enduring deficits in mobility and posture owing to non-progressive injury to the infant or developing brain. CP is the predominant etiology of physical impairment observed in children. Research indicates a global prevalence of 1.6 per 1,000 live births in developing nations and 3.4 per 1,000 in low- and middle-income countries. Ninety percent of all CP patients demonstrate spasticity as a symptom. Spasticity is characterized by a speed-dependent augmentation of excessive stretch reflexes, stemming from the hyperexcitability of these reflexes due to upper motor neuron injury. Management of spasticity includes physical therapy techniques, antispasmodic medication, botulinum toxin administration, orthotic devices, therapeutic exercises, and surgical interventions. Stretching exercises constitute one of the initial therapeutic interventions and have been employed for numerous years. Certain studies indicate that the impact of conventional stretching on joint range of motion and spasticity is constrained. If spasticity is not appropriately managed, it may hinder motor learning and the development of movement abilities, leading to various functional impairments such as joint contractures and gait issues over time, while also causing changes in muscle architecture. Muscle architecture denotes the configuration of fibers or fascicle bundles within the muscle. It encompasses the fascicle length and pennation angle.

The length of a muscle fiber or fascicle correlates with the muscle's maximal excursion and contraction velocity, reflecting the number of sarcomeres arranged in series. The physiological cross-sectional size of a muscle is directly related to its maximum force production capability and the quantity of sarcomeres arranged in parallel. Numerous investigations have documented a reduction in fascicle length in the afflicted limbs of children with cerebral palsy. The extension of fascicle length can beneficially impact children's functional capabilities by improving the muscle's length-tension and force-velocity properties. Consequently, the extension of fascicle length is crucial for enhancing children's motor functions and functional capabilities. Ultrasonography of the musculoskeletal system serves as a potential instrument for assessing alterations in in vivo muscle architecture. It has been utilized in numerous research studies, including the pediatric population, to elucidate muscle anatomy. One study indicated that high-speed passive stretching may enhance muscle fascicle length in spastic muscles.

The hypothesis of the study is that rapid stretching exercises administered to children with cerebral palsy who have undergone BoNT-A treatment will yield superior outcomes in spasticity, functional status, and muscle architecture compared to conventional speed stretching.

Method:

Study Design and Participants:

The present study is designed as a prospective, single-blind, randomized controlled trial. It investigates the effects of high-velocity and standard ankle stretching exercises, added to a standard physical therapy program, on functional status, muscle architecture, and spasticity in children with cerebral palsy. Furthermore, it evaluates the contribution of these parameters to gait. The minimum required number of extremities per group was calculated as 23. Considering a 10% potential dropout rate, 26 extremities (17 children) per group were allocated. Accordingly, a total of 52 extremities from 34 children aged between 2 and 8 years were planned for inclusion.

All participants receive botulinum toxin-A (BoNT-A) injections into the gastrocnemius muscle in accordance with clinical indications and the guidelines of the Health Implementation Communiqué (SUT). Participants scheduled for BoNT-A injections and presenting to the Physical Medicine and Rehabilitation outpatient clinic of Erciyes University Faculty of Medicine undergo standardized clinical history, physical examination, anthropometric measurements, observational gait analysis, and ultrasound assessments.

Following BoNT-A administration, all participants undergo a standardized physical therapy and rehabilitation program delivered by the same physiotherapist three times a week for four weeks. The intervention group receives a high-velocity passive stretching protocol, while the control group follows a standard stretching protocol. Treatment protocols are explained to families during the hospital-based therapy period to ensure accurate implementation.

After completing the four-week in-hospital therapy, all participants continue with a home-based exercise program until the 6th month. These exercises are performed by families and are designed to replicate the stretching routines taught during hospital sessions, particularly in terms of velocity and technique. Adherence to the home program is monitored through telephone follow-ups at the 2nd, 4th, and 5th months.

Participants are randomly assigned to either the high-velocity stretching or standard stretching protocol group, both combined with the standardized physical therapy regimen. Assessments are conducted at baseline (pre-injection) and at the 1st, 3rd, and 6th months post-injection. The eligibility criteria and detailed participant selection process are described in the Eligibility section.

Randomization:

Participants will be assigned to intervention and control groups using stratified randomization based on GMFCS staging. The website "https://www.randomizer.org/" will be used for the randomization process. The randomization procedure will be conducted by an independent research assistant who will store the randomization codes and will not be involved in the study process. The evaluator will be completely blinded to group assignments and will have no information regarding the treatment process. The physiotherapist administering the treatment will not be blinded to the treatment methods but will not participate in the evaluation stages. This approach ensures impartiality in randomization and evaluation processes.

Interventions:

• Standard Rehabilitation Protocol: Participants in both groups undergo a one-hour physical therapy program including strengthening exercises, weight-bearing, balance, proprioception, and walking training.

• Stretching Protocol: Stretching will be applied in the same position for participants in both groups. Participants lie supine on a foam mat, and the physiotherapist positions beside the participant, opposite the leg to be stretched. The starting position for stretching is achieved by lifting the leg to 90° knee flexion. To stretch the gastrocnemius muscle, the physiotherapist's hand is placed flat on the foot with a smartphone fixed around the heel and the palm flat against the foot. The knee is supported and brought into full extension, with pressure applied to the proximal tibia for stabilization. Once the knee is locked in full extension, the ankle is dorsiflexed, and pressure is applied to the plantar surface, stretching the muscle until maximum dorsiflexion is reached. Standardization for both groups is provided using smartphone applications. The metronome app standardizes start, end, and rest intervals. Speed measurements are standardized using the Phyphox application. Angular velocity data taken with a smartphone fixed to the plantar region of the foot are transferred to an Excel file. The data are in radians/sec and will be converted to degrees/sec in Excel.

In the intervention group, stretching starts as described above, first at a slow speed (V1) for 5 minutes, followed by fast stretching (V3) for 10 minutes (to induce the catch sensation), as per Tardieu's method. A 1-minute rest period is provided after each stretch. This protocol is performed three times a week for four weeks under physiotherapist supervision, after which families continue the exercises as home exercises without speed measurements for up to 6 months. In the control group, standard stretching is applied with 10 repetitions of 60 seconds and 30 seconds of rest intervals for each leg, three times a week for a total of 15 minutes per session. Similarly, families continue exercises at home for 6 months after the 4-week period.

Outcome Measures:

Detailed in the Outcome Measurements section.

Power Analysis:

Sample size was determined using G*Power software (version 3.1.9.7), based on Kavano et al.'s study. Their study found that 12 weeks after botulinum toxin injections to the gastrocnemius, fascicle length increased by approximately 6% (at rest) and 14% (at maximum dorsiflexion). Assuming a similar difference in fascicle length between intervention and control groups in the current study, with a standard deviation of 3.6, 80% power, and a Type I error of 0.05, at least 23 limbs per group were calculated as necessary. Considering a 10% dropout rate, 26 limbs per group (17 children) were planned, totaling 34 patients.

Statistical Analysis:

All statistical analyses will be conducted using SPSS version 22.0. Normality of the data will be tested using the Shapiro-Wilk test. Baseline (pre-intervention) numerical data from both groups will be compared using independent samples t-tests (if normally distributed) or Mann-Whitney U tests (if not normally distributed). Primary (fascicle length) and secondary outcomes (pennation angle, muscle thickness, spasticity scores, OGA scores, GMFM-66 scores, and ROM scores) will be analyzed for intra-group and inter-group (intervention vs. control) differences across different time points (pre-treatment, post-treatment at 1 month, 3 months, and 6 months) using repeated measures mixed-model ANOVA. Bonferroni correction will be applied to determine specific time points of significant differences. Linear regression analysis will assess the relationship between changes in fascicle length and independent variables (group, time, spasticity score, etc.). Chi-square or Fisher's exact tests will be used for categorical variables. A significance level of p<0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 8 years diagnosed with cerebral palsy of the hemiplegic or diplegic type according to the Rosenbaum criteria
* Presence of spasticity in the ankle plantar flexors with a Modified Ashworth Scale (MAS) score of 1, 1+, 2, or 3, and a clinical indication for BoNT-A injection into the gastrocnemius or gastrocnemius/soleus muscles at this stage of treatment
* Gross Motor Function Classification System (GMFCS) levels of 1, 2, or 3 (ambulatory)

Exclusion Criteria:

* Having a neuromuscular disorder other than cerebral palsy
* Presence of a fixed foot deformity
* Receiving serial casting or spasticity treatments (e.g., baclofen or BoNT-A) within the past 6 months
* History of surgery
* Having intellectual or behavioral difficulties, or comorbid conditions (such as cardiac, respiratory disorders or uncontrolled seizures) that prevent safe participation in exercise

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Fascicle length measured via ultrasound in maximum dorsiflexion and resting positions. | Patients will be assessed at the hospital before the BoNT-A injection and at the 1st, 3rd, and 6th months following the injection
  The patient will be positioned prone with the ankle hanging freely off the edge of the examination table. Imaging will be performed over the medial gastrocnemius in full knee extension (0° flexion) during both maximum dorsiflexion (MDF) and resting positions. Using two-dimensional ultrasound, the length of the longest fascicle extending between the superficial and deep fascia will be measured at the thickest point of the medial gastrocnemius muscle.

SECONDARY OUTCOMES:
Pennation angle | Patients will be assessed at the hospital before the BoNT-A injection and at the 1st, 3rd, and 6th months following the injection
  The patient will be positioned prone with the ankle hanging freely off the edge of the examination table. Imaging will be performed over the medial gastrocnemius in full knee extension (0° flexion) during both maximum dorsiflexion (MDF) and resting positions. Using two-dimensional ultrasound, fascicles extending between the superficial and deep fascia at the thickest point of the medial gastrocnemius muscle will be selected.. The pennation angle will be measured as the angle formed between the orientation of the muscle fascicles and the superficial fascia (representing the line of action of the tendon)
Gastrocnemius muscle thickness | Patients will be assessed at the hospital before the BoNT-A injection and at the 1st, 3rd, and 6th months following the injection
  The thickness of the medial gastrocnemius muscle was measured at its thickest point using two-dimensional (2D) B-mode ultrasound imaging. The measurement was defined as the maximum perpendicular distance between the superficial and deep fasciae of the muscle, as seen in a transverse ultrasound image. Measurements were performed in two different ankle joint positions, both with the knee fully extended: (1) at rest, and (2) at maximum dorsiflexion, achieved by manually moving the ankle to the end of its range of motion in the sagittal plane.
Assessment of Spasticity (Modifiye ashworth classification) | Patients will be assessed at the hospital before the BoNT-A injection and at the 1st, 3rd, and 6th months following the injection
  Muscle tone was evaluated using the Modified Ashworth Scale (MAS), a widely used six-point ordinal scale ranging from 0 to 4, where higher scores indicate increased spasticity. The assessment was performed by a clinician who passively moved the target limb rapidly through its full available range of motion while evaluating the resistance felt during the movement. In this study, a MAS score of 1+ was converted to a value of 2 for statistical analysis. Subsequently, MAS scores of 2, 3, and 4 were recoded as 3, 4, and 5, respectively, in order to provide a linearized scale for comparative purposes.
Assessment of Spasticity (Tardie Scale) | Patients will be assessed at the hospital before the BoNT-A injection and at the 1st, 3rd, and 6th months following the injection
  Spasticity of the ankle plantar flexor muscles was assessed using the Tardieu Scale, which evaluates the muscle response to passive stretching at different velocities. Two standardized velocities were applied: V1 (as slow as possible) and V3 (as fast as possible). For each muscle, both the angle of muscle reaction (R1) and the full passive range of motion (R2) were measured using a standard plastic goniometer. Assessments were conducted for the gastrocnemius (with the knee fully extended) and the soleus (with the knee flexed at 90°). The neutral ankle joint position was defined as 0°, with dorsiflexion recorded as positive and plantar flexion as negative values.
  The dynamic component of spasticity was quantified by calculating the difference between R2 and R1 (R2-R1), which reflects the velocity-dependent resistance of the muscle. Greater R2-R1 values indicate increased dynamic spasticity, which is considered a negative outcome. In addition to angle measurements, the muscle reaction
Range of Motion | Patients will be assessed at the hospital before the BoNT-A injection and at the 1st, 3rd, and 6th months following the injection
  The researcher will measure the patient's maximal dorsiflexion and maximum plantar flexion angles using a plastic goniometer with the knee fully extended.
Observational Gait Analysis | Patients will be assessed at the hospital before the BoNT-A injection and at the 1st, 3rd, and 6th months following the injection
  A measurement instrument employed to evaluate ambulation capabilities in children. It enables observers to assess children's walking via video recordings and rate them according to parameters such as ankle and knee positioning
The Gross Motor Function Measure-66 | Patients were assessed at the hospital before the BoNT-A injection and at the 1st, 3rd, and 6th months after the injection.
  GMFM-66 has five domains: A - Lying and Rolling, B - Sitting, C - Crawling and Kneeling, D - Standing and Walking, and E - Running and Jumping. This is the definitive scale for assessing the motor functions of a kid with cerebral palsy. The GMFM-66 version was created following the Rasch analyses, which entailed the elimination of 66 items from the GMFM-88. The Turkish translation will be utilized in our investigation

CONTACTS AND LOCATIONS:
Overall Officials: İsa C Associate Professor, Principal Investigator — Erciyes University Faculty of Medicine Hospital
Locations (1):
- Erciyes University Faculty of Medicine Hospital, Kayseri, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All participants' demographic and research data (i.e. outcome measures) are recorded in detail. They will be shared if requested by ICMJE or other legal authorities.

REFERENCES:
- [Background] Lichtwark GA, Bougoulias K, Wilson AM. Muscle fascicle and series elastic element length changes along the length of the human gastrocnemius during walking and running. J Biomech. 2007;40(1):157-64. doi: 10.1016/j.jbiomech.2005.10.035. Epub 2005 Dec 20. PMID 16364330
- [Background] Benard MR, Becher JG, Harlaar J, Huijing PA, Jaspers RT. Anatomical information is needed in ultrasound imaging of muscle to avoid potentially substantial errors in measurement of muscle geometry. Muscle Nerve. 2009 May;39(5):652-65. doi: 10.1002/mus.21287. PMID 19291798
- [Background] Gracies JM, Burke K, Clegg NJ, Browne R, Rushing C, Fehlings D, Matthews D, Tilton A, Delgado MR. Reliability of the Tardieu Scale for assessing spasticity in children with cerebral palsy. Arch Phys Med Rehabil. 2010 Mar;91(3):421-8. doi: 10.1016/j.apmr.2009.11.017. PMID 20298834
- [Background] Zurawski E, Behm K, Dunlap C, Koo J, Ismail F, Boulias C, Reid S, Phadke CP. Interrater Reliability of the Modified Ashworth Scale with Standardized Movement Speeds: A Pilot Study. Physiother Can. 2019 Fall;71(4):348-354. doi: 10.3138/ptc-2018-0086. PMID 31762545
- [Background] Theis N, Korff T, Mohagheghi AA. Does long-term passive stretching alter muscle-tendon unit mechanics in children with spastic cerebral palsy? Clin Biomech (Bristol). 2015 Dec;30(10):1071-6. doi: 10.1016/j.clinbiomech.2015.09.004. Epub 2015 Sep 8. PMID 26403361
- [Background] Banky M, Clark RA, Mentiplay BF, Olver JH, Kahn MB, Williams G. Toward Accurate Clinical Spasticity Assessment: Validation of Movement Speed and Joint Angle Assessments Using Smartphones and Camera Tracking. Arch Phys Med Rehabil. 2019 Aug;100(8):1482-1491. doi: 10.1016/j.apmr.2018.11.026. Epub 2019 Jan 24. PMID 30684484
- [Background] Kawano A, Yanagizono T, Kadouchi I, Umezaki T, Chosa E. Ultrasonographic evaluation of changes in the muscle architecture of the gastrocnemius with botulinum toxin treatment for lower extremity spasticity in children with cerebral palsy. J Orthop Sci. 2018 Mar;23(2):389-393. doi: 10.1016/j.jos.2017.10.012. Epub 2017 Nov 14. PMID 29146092
- [Background] Davis JF, Khan T, Thornton M, Reeves ND, DeLuca M, Mohagheghi AA. High Velocity Passive Stretching Mimics Eccentric Exercise in Cerebral Palsy and May Be Used to Increase Spastic Muscle Fascicle Length. Bioengineering (Basel). 2024 Jun 13;11(6):608. doi: 10.3390/bioengineering11060608. PMID 38927844